CLINICAL TRIAL: NCT07349849
Title: Exploratory Study on mRNA Therapeutic Drug Targeting CD19 for the Treatment of Hematologic Malignancies
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Xi Zhang, MD, Professor, Xinqiao Hospital of Chongqing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: in vivo CAR-T of CD19
Record Dates: First submitted 2025-12-19; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: B-cell Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- in vivo CAR-T drug based on LNP-mRNA (Experimental)
  Interventions: Drug: in vivo CAR-T drug based on LNP-mRNA

INTERVENTIONS:
Drug: in vivo CAR-T drug based on LNP-mRNA — in vivo CAR-T drug based on LNP-mRNA

SUMMARY:
Malignant hematological tumors mainly derived from adult B cells are mainly acute lymphoblastic leukemia (ALL) and non Hodgkin lymphoma (NHL). Overall, although existing therapies have significantly improved the survival rates of most patients, the treatment of relapsed/refractory patients still faces significant challenges. CD19 is one of the most clinically valuable targets for B-cell malignant hematological tumors.

The advent of COVID-19 vaccine has brought LNP mRNA technology into the public's view. After years of development, it not only shines brilliantly in COVID-19 vaccine, but also is widely used in the treatment and exploration of cancer, rare diseases and other fields. Lipid nanoparticles (LNP) are currently the most mature non viral delivery platform, capable of protecting mRNA from nuclease degradation, promoting intracellular uptake, and achieving efficient translation in vivo.

The core of LNP-mRNA technology targeting CD19 is to encapsulate the mRNA encoding specific proteins (such as anti-CD19 related proteins) in lipid nanoparticles and deliver them to the body through intravenous or intramuscular injection.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age range of 18-70 years old, gender not limited;
* 2. Expected survival time exceeds 12 weeks;
* 3. B-cell lymphoma or lymphocytic leukemia diagnosed with CD19+, with no standard treatment options recommended according to guidelines
* 4. There are assessable lesions (applicable only to lymphoma patients);
* 5. The physical fitness status score of the Eastern Cancer Collaboration Group (ECOG) is 0 or 1;
* May involve other inclusion criteria

Exclusion Criteria:

* 1. Accompanied by other uncontrolled malignant tumors;
* 2. Previously received chimeric antigen receptor therapy or other transgenic T cell therapy;
* 3. Known history of HIV or hepatitis B (HBsAg positive and HBV DNA reaching the detection limit) or hepatitis C virus (anti HCV positive) infection;
* 4. Participants with a history of CNS lymphoma, malignant cells in cerebrospinal fluid, or brain metastases;
* 5. The researcher believes that there are any other factors that are not suitable for the study participants to enter this trial.

May involve other exclusion criteria

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) and its incidence rate | Within 28 days after the initial treatment
Maximum tolerated dose (MTD) or optimal biological dose (OBD) | 3 months

SECONDARY OUTCOMES:
Objective response rate (ORR) | 1 month
Disease control rate (DCR) | Through study completion, an average of 2 years
Progression free survival (PFS) | From date of initial treatment until the date of first comfired progression or date of death from any cause, whichever came first, assessed up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hematology, Xinqiao Hospital, Chongqing, Chongqing Municipality, China